CLINICAL TRIAL: NCT06053970
Title: Prospective, Randomized, Exploratory Study Evaluating the Effect of Moving Virtual Scenes on Postural Balance in a Subacute Stroke Rehabilitation Setting
Brief Title: Study Evaluating the Effect of Moving Virtual Scenes on Postural Balance in a Stroke Rehabilitation Setting
Acronym: VR-REACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: FondationbHopale (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HOP23-RIPH2-10
Record Dates: First submitted 2023-08-30; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-07

CONDITIONS: Stroke Rehabilitation; Postural Equilibrium

STUDY DESIGN:
Intervention Model Description: Recruitment of twenty patients. The order of the virtual reality scenes will be randomly selected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Random order of virtual scenes (Other): Eight measurements on a stabilometry platform will be performed for each of the VR signals, in random order:
  Signal A Direction: anteroposterior Speed: 5 m/s
  Signal B Direction: anterior-posterior Speed: 5 m/s
  Signal C Direction: Oblique forward and downward Speed: 5 m/s
  Signal D Direction: Oblique forwards and upwards Speed: 5 m/s
  Signal E Direction: Oblique forwards and to the right Speed: 5 m/s
  Signal F Direction: Oblique forward and left Speed: 5 m/s
  Signal G Direction: antero-posterior + Clockwise tunnel rotation at 10°/s Speed: 5 m/s
  Signal H Direction: antero-posterior + Counter-clockwise tunnel rotation at 10°/s Speed: 5 m/s
  Interventions: Other: Assessing postural responses induced by visual stimulation (Visual Evoked postural responses, VEPR)

INTERVENTIONS:
Other: Assessing postural responses induced by visual stimulation (Visual Evoked postural responses, VEPR) — The intervention will last 60 minutes and will include an assessment of the Berg Balance Scale (BBS), the collection of stabilometric data, the collection of the numerical difficulty scale, the Fast Motion Sickness Scale (FMS) and will end with a break after exposure to VR.
  The various conditions will be carried out in this order:
  * Eyes open with VR headset simulating a static environment
  * Eyes closed with VR helmet off
  * Eight measurements on a stabilometry platform will be taken for each of the VR signals, in random order

SUMMARY:
This is an interventional, prospective, randomized, monocentric study designed to develop medical knowledge.

Virtual reality is increasingly used in rehabilitation. The aim of virtual reality is to investigate motor interactions in a fictitious, configurable environment, in order to train specific functions and transpose improvements into everyday life.

The main objective of this study is to investigate the influence of different moving virtual scenes on the general spatiotemporal parameters of pressure centers, in a sub-acute stroke rehabilitation context.

This would help health professionals to assess the most suitable VR exercise in function of patient's difficulties.

During this study, patient movements while viewing 8 different virtual reality scenes will be recorded using a motion platform during a single session.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18
* Adult patient in rehabilitation stay (day or full hospitalization) following a first stroke less than 6 months old.
* One of the rehabilitation objectives is to improve balance
* Ability to understand exercise instructions
* Ability to stand for at least one minute with eyes closed, safely and without technical assistance
* Ability to walk at least with technical assistance and/or supervision
* Patient having given their informed consent
* Patient affiliated to a social security scheme

Non -inclusion criteria :

* Patients with epilepsy, controlled or not
* Patients undergoing rehabilitation following a stroke in the posterior fossa
* Known history of vestibular or cerebellar balance disorders
* Patients with orthopedic or traumatological impairment preventing stabilometric measurement on a force platform without footwear
* Patient under legal protection measure
* Severe phasic disorders that may prevent the expression of the will to stop viewing virtual scenes or to respond to numerical scales
* Pregnant or breastfeeding woman
* Known history of motion sickness
* Patient participating or having participated in the balance rehabilitation program with virtual reality within the rehabilitation center during their stay

Exclusion Criteria :

* Cyberkinetosis represented by a score greater than or equal to 15 on the Fast Motion Sickness scale
* Poor tolerance for wearing a virtual reality headset
* Significant visual impairment preventing the perception of the stimulus visual

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Total length of pressure center displacement (in mm) | During the procedure (virtual reality session).
  Length of pressure will be recorded on a force platform under different conditions:
  * Eyes open with VR headset simulating a static environment
  * Eyes closed with VR helmet off
  * In 8 VR conditions simulating movement (in random order)
Displacement speed of the center of pressure (in mm.s-1) | During the procedure (virtual reality session).
  Displacement speed of the center of pressure will be recorded on a force platform under different conditions:
  * Eyes open with VR headset simulating a static environment
  * Eyes closed with VR helmet off
  * In 8 VR conditions simulating movement (in random order)

CONTACTS AND LOCATIONS:
Locations (1):
- FONDATION HOPALE - Centre de rééducation Ste Barbe, Fouquières-lès-Lens, France